CLINICAL TRIAL: NCT01371201
Title: First International Randomized Study in Malignant Progressive Pheochromocytoma and Paraganglioma (PPGL)
Brief Title: First International Randomized Study in Malignant Progressive Pheochromocytoma and Paraganglioma
Acronym: FIRSTMAPPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); European Network for the Study of Adrenal Tumours (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGR2010/1715; 2010-024621-20 (EudraCT Number); MSI/A110356-31 (Other: AFSSAPS)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Malignant Progressive Pheochromocytoma and Paraganglioma (PPGL)
MeSH Terms: conditions — Paraganglioma | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib (Experimental): sunitinib 37.5 mg per day
  Interventions: Drug: Sunitinib
- Placebo (Placebo Comparator): Placebo 37.5 mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sunitinib — sunitinib 37.5 mg per day
  Other Names: Sutent
  Arms: Sunitinib
Drug: Placebo — Placebo 37.5 mg per day
  Arms: Placebo

SUMMARY:
The FIRSTMAPPP study is a randomized, double-blind, phase II, international, multicenter study which aims to determine the efficacy of Sunitinib on the progression-free survival at 12 months in subjects with progressive malignant pheochromocytoma and paraganglioma treated with sunitinib at a starting dose of 37.5 mg daily (continuous dosing).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the efficacy of Sunitinib on the progression-free survival at 12 months in subjects with progressive malignant pheochromocytoma and paraganglioma treated with sunitinib at a starting dose of 37.5 mg daily (continuous dosing).

SECONDARY OBJECTIVES:

* To determine overall survival and progression free survival.
* To determine time to progression.
* To determine objective response rate at one year.
* To determine time to and duration of tumor response.
* To assess safety profile including a dedicated cardiovascular management (home-blood pressure monitoring, ECG and echocardiography).

EXPLORATORY OBJECTIVES:

-Identification of predictors of response as well as surrogate markers of overall survival is anticipated

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant PPGL, based on imaging or biopsy evidence of metastases in liver, bones, lungs and or lymph nodes, combined with at least one of two further confirmatory diagnoses: 1. diagnosis of PPGL from histopathological review of resected or biopsied tissue performed by a skilled pathologist (centralized review will be performed in all cases either before enrolment in case of any doubt or during the study); or 2. in patients where tumor tissue is unavailable for formal pathological review, from combined biochemical and functional imaging evidence of PPGL (e.g., MIBG scintigraphy combined with consistently and highly elevated plasma or urine levels of metanephrines).
* Metastatic disease not amenable to surgical resection
* Pre-treated or not
* Whatever the genetic status (sporadic or inherited)
* Evaluable disease according to RECIST 1.1 criteria
* Progressing disease within 18 months at imaging prior to randomization according to RECIST. The recent scan indicating progression may be used as the screening scan if within 28 days of randomization
* ECOG performance status 0-2
* Life expectancy ≥ 6 months as prognosticated by the physician
* Age ≥18 years, no superior limit
* Adequate bone marrow reserve (Hb > 8, neutrophils ≥ 1500/mm³ and platelets ≥80.000/mm³)
* Effective contraception in pre-menopausal female and male patients
* Negative pregnancy test
* Patient´s signed written informed consent
* Ability to comply with the protocol procedures
* Ability to take oral medication

Exclusion Criteria:

* Large or small cell-poorly differentiated neuroendocrine carcinoma according to WHO 2000 classification
* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
* Severe renal (GFR <30ml/mn or nephrotic syndrome) or hepatic insufficiency (ALT / AST > 2.5 x ULN or ALT/AST >5 x ULN if liver function abnormalities are due to the underlying malignancy and/or total serum bilirubin > 2.5 x ULN)
* Patients with cardiac events within the previous 12 months, such as myocardial infarction (including severe/unstable angina pectoris), coronary/peripheral artery bypass graft, revascularization procedure symptomatic congestive heart failure (CHF, ejection fraction <45%), ), uncontrolled cardiac arrhythmia, clinically significant bradycardia, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Hypertension that cannot be controlled despite medications (>=160/95 mmHg despite optimal medical therapy)
* Abnormal cardiac function with 12 lead ECG. Ongoing cardiac dysrhythmias of NCI CTC grade >=2, atrial fibrillation of any grade, or prolongation of the QTc interval to >470 msec for males or >480 msec for females.
* Brain metastases (exception if stable and asymptomatic for more than 3 months)
* Pregnancy or breast feeding
* Previous treatment with the drug under study. Prior systemic treatment with any tyrosine kinase inhibitors or anti VEGF angiogenic inhibitors.
* Current treatment with another investigational drug.
* Treatment with potent CYP3A4 inhibitors and inducers within 7 and 12 days, respectively prior to study drug administration
* Concomitant treatment with therapeutic doses of anticoagulants. Low dose warfarin (Coumadin) up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed as well as heparin-based anticoagulation
* Prior treatments with chemotherapy, immunotherapy, somatostatine analog therapy drug , thoracic radiotherapy within 4 weeks prior to inclusion
* Major surgery for any cause or local radiotherapy within one month prior to visit 1
* Liver embolisation therapy within the last 3 months prior visit 1 except if progression is demonstrated and embolised lesion not used as targets
* Unrecovered toxicity from any kind of therapy
* Active or suspected acute or chronic uncontrolled disease that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-12-22 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 12 months | 12 months
  Progression will be assessed by RECIST 1.1 performed every 3 months (centralized imaging)

SECONDARY OUTCOMES:
Objective Response Rates (ORR) | 12 months
Duration of response (DR) | 12 months
Overall Time to Progression (TTP) | 12 months
Overall survival (OS) | 12 months
Number of Adverse Events assessed using NCI -CTC V4 criteria | 12 months
  Number and description of adverse events and number of patients with adverse events according to NCI -CTC V4 criteria
Number of patients with cardiovascular toxicity tolerance assessed by specific organisation for blood pressure monitoring | 12 months
  Cardiovascular tolerance will be assessed by specific organisation for blood pressure monitoring
Bone Pain evaluation on the Visual Analog Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Baudin, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- Institut de Cancérologie Gustave roussy, Villejuif, France
- Universitätsklinikum Würzburg, Würburg, Germany
- University of Padova, Padua, Italy
- Radboud University Nijmegen Medical Centre, Nijmegen, GA, Netherlands

REFERENCES:
- [Derived] Baudin E, Goichot B, Berruti A, Hadoux J, Moalla S, Laboureau S, Nolting S, de la Fouchardiere C, Kienitz T, Deutschbein T, Zovato S, Amar L, Haissaguerre M, Timmers H, Niccoli P, Faggiano A, Angokai M, Lamartina L, Luca F, Cosentini D, Hahner S, Beuschlein F, Attard M, Texier M, Fassnacht M; ENDOCAN-COMETE; ENSAT Networks. Sunitinib for metastatic progressive phaeochromocytomas and paragangliomas: results from FIRSTMAPPP, an academic, multicentre, international, randomised, placebo-controlled, double-blind, phase 2 trial. Lancet. 2024 Mar 16;403(10431):1061-1070. doi: 10.1016/S0140-6736(23)02554-0. Epub 2024 Feb 22. PMID 38402886
- [Derived] Fankhauser M, Bechmann N, Lauseker M, Goncalves J, Favier J, Klink B, William D, Gieldon L, Maurer J, Spottl G, Rank P, Knosel T, Orth M, Ziegler CG, Aristizabal Prada ET, Rubinstein G, Fassnacht M, Spitzweg C, Grossman AB, Pacak K, Beuschlein F, Bornstein SR, Eisenhofer G, Auernhammer CJ, Reincke M, Nolting S. Synergistic Highly Potent Targeted Drug Combinations in Different Pheochromocytoma Models Including Human Tumor Cultures. Endocrinology. 2019 Nov 1;160(11):2600-2617. doi: 10.1210/en.2019-00410. PMID 31322702
- See also: Sponsor website — http://www.igr.fr/